CLINICAL TRIAL: NCT03656354
Title: Identification of Heart Failure Patients by Seismocardiography; a Comparison With Echocardiography and Brain Natriuretic Peptide
Brief Title: Identification of Heart Failure Patients by Seismocardiography
Acronym: SCG-HF
Status: Completed | Type: Observational
Sponsor: Acarix (Industry)
Responsible Party: Sponsor
Other Study IDs: AC013AOU
Record Dates: First submitted 2018-06-27; First posted 2018-09-04 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
Keywords: seismocardiography
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Seismocardiography — Seismocardiography recording

SUMMARY:
The aim of the current study is to develop and validate an algorithm based on seismocardiography recordings to detect heart failure. Echocardiography will be used as the golden standard for defining patients with heart failure.

DETAILED DESCRIPTION:
Seismocardiography is inspired from methods for the analysis of seismic activity and can be used to describe the heart's movements using a specially developed sensor placed on the patient's chest. The project aims to describe the motion of the heart using automated computer analysis of the seismocardiography signal for development of a simple method for the analysis of myocardial performance.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or older
* Clinically suspected heart failure, and referred to an outpatient clinic
* Be able and willing to comply with the clinical investigational plan
* Have signed the informed consent form

Exclusion Criteria:

* Known HF
* Known atrial fibrillation
* Acute coronary syndrome
* Implanted donor heart, mechanical heart, mechanical heart pump, pacemaker or Cardioverter Defibrillator (ICD)
* Implanted electronic equipment in the area above and around the heart
* Significant operation scars, abnormal body shape, fragile or compromised skin in the seismocardiographic recording area (fourth left Inter Costal space and xiphoid process)
* Pregnancy

Extension study:

Inclusion criteria

1. Male or female, aged 18 years or older
2. Newly diagnosed HFREF
3. Be able and willing to comply with the clinical investigational plan
4. Have signed the informed consent form

Exclusion criteria

1. Known atrial fibrillation
2. Acute coronary syndrome
3. Implanted donor heart, mechanical heart, mechanical heart pump, pacemaker or Cardioverter Defibrillator (ICD)
4. Implanted electronic equipment in the area above and around the heart
5. Significant operation scars, abnormal body shape, fragile or compromised skin in the seismocardiographic recording area (fourth left Inter Costal space and xiphoid process)
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically suspected heart failure
  Extension study:
  Patients with newly diagnosed HFrEF
Sampling Method: Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Area under the receiver-operator characteristic curve, sensitivity, specificity, and positive and negative predictive value of seismocardiography in detection of heart failure. | 1 day
  Heart failure defined as heart failure with reduced ejection fraction, heart failure with mid-range ejection fraction and heart failure with preserved ejection fraction combined.

SECONDARY OUTCOMES:
Area under the receiver-operator characteristic curve, sensitivity, specificity, and positive and negative predictive value of seismocardiography and NT-proBNP, respectively, in detection of heart failure with reduced ejection fraction | 1 day
Area under the receiver-operator characteristic curve, sensitivity, specificity, and positive and negative predictive value of seismocardiography in detection of heart failure with mid-range ejection fraction. | 1 day
Area under the receiver-operator characteristic curve, sensitivity, specificity, and positive and negative predictive value of seismocardiography in detection of heart failure with preserved ejection fraction. | 1 day
Adverse events related to the CADScor seismo device. | 1 day
  Count of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Peter Søgaard, MD, DMSc, Principal Investigator — Aalborg University Hospital; Jacob Møller, MD, DMSc, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No